CLINICAL TRIAL: NCT06138574
Title: Effects of Dexmetomidine and Remifentanil Used for Controlled Hypotension in Septorhinoplasty Surgery on Cardiac Electrophysiology: Prospective Randomized Study
Acronym: Effects of Dex
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Saglik Bilimleri Universitesi Gazi Yasargil Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Hülya Tosun Söner, HTosunSoner, Saglik Bilimleri Universitesi Gazi Yasargil Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HTosun
Record Dates: First submitted 2023-11-14; First posted 2023-11-18 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Rhinoplasty Surgery
MeSH Terms: interventions — Dexmedetomidine; Remifentanil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Effects of Dexmetomidine (Active Comparator): Patients in this group will be given dexmedetomidine infusion during the intraoperative period to provide controlled hypotension.
  Interventions: Drug: Dexmedetomidine
- Effects of Remifentanil (Active Comparator): Patients in this group will be given remifentanil infusion during the intraoperative period to provide controlled hypotension.
  Interventions: Drug: Remifentanil

INTERVENTIONS:
Drug: Dexmedetomidine — After the induction of general anesthesia, one group (Group: 1) will be administered dexmedotomidin infizyon and group (Group :2)remifentanil
  Arms: Effects of Dexmetomidine
Drug: Remifentanil — Remifentanil
  Arms: Effects of Remifentanil

SUMMARY:
Our aim in this treatment was to reveal the effects of remifentanil and dexmetomidine, which we used to provide controlled hypotension in septorhinoplasty surgery, on cardiac electrophysiology. We planned to compare the patients by recording preoperative and postoperative ECGs. We also planned to record the patients' intraoperative blood pressure, saturation, and pulse rate, rickeragitation scale, and vas score.

ELIGIBILITY:
Inclusion Criteria:

* patients with an ASA score of I and between the ages of 17-45 years, who were to undergo general anesthesia with sevofulurane were included in the study.

Exclusion Criteria:

Patients aged <17 and >45 years, patients with liver and/or kidney failure, obese patients (BMI >30), trauma patients, ASA II-III-IV patients, patients with bleeding disorders, those using drugs that may affect the coagulation system, patients with cardiomyopathy, cerebrovascular disease, immobility, and malnutrition were excluded from the study.

-

Ages: 17 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 72 (Estimated)
Dates: Start 2023-12-01 (Estimated); Primary Completion 2024-02-01 (Estimated); Study Completion 2024-03-30 (Estimated)

PRIMARY OUTCOMES:
iceb | preoperative and postoperative (immediatly after extubation)
  Qt\Qrs

SECONDARY OUTCOMES:
Riker Agitation Scale | Immediately after extubation
  7 -Dangerous Agitation, 6 - Very Agitated, 5 - Agitated, 4 - Calm and Cooperative, 3 - sedated, 2- Very Sedated, 1 -Unarousable
mean arterial pressure | when you come to the operating room table after anesthesia induction Intraoperative 30 minutes after extubasion
  mmHg
heart rate | when you come to the operating room table after anesthesia induction Intraoperative 30 minutes after extubasion
  beats\minute
Numeric Rating Scale | Postoperative 0-2 hours
  They will be numbered from 1 to 10. 1 mildest 10 most severe pain